CLINICAL TRIAL: NCT06480266
Title: Influence of Protein Intake on Muscle Mass and Health-related Quality of Life During and After Radiotherapy in Patients With Various Tumor Diseases
Brief Title: Influence of Protein Intake on Muscle Mass and Health-related Quality of Life During and After Radiotherapy
Acronym: pROtein
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Franziska Hausmann, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA1/101/23
Record Dates: First submitted 2024-02-06; First posted 2024-06-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Malnutrition; Cachexia
Keywords: Cancer; Radiotherapy; Nutrition; Sarcopenia; Inflammation; Microbiome
MeSH Terms: conditions — Malnutrition; Cachexia; Neoplasms; Sarcopenia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The influence of radiotherapy on the protein intake and muscle mass of patients has not been extensively investigated to date. It is also unclear whether the localization of the tumor disease and thus the radiation field have different effects. Therefore, with the pilot study presented here, we would like to record the nutritional uptake of patients before and after radiotherapy. The aim is to determine the amount of energy and protein intake as well as the timing of protein intake. Furthermore, the relationship between the timing of protein intake and muscle mass will be investigated.

DETAILED DESCRIPTION:
Many studies have shown that cancer patients have a very high prevalence of malnutrition. Several large-scale studies have reported that 50-80% of these patients are affected by involuntary weight loss, with the extent of weight loss depending on the tumor location and the type and stage of the disease. It has been widely reported that nutritional interventions are essential in cancer patients. Nevertheless, nutritional support is still not universally accessible to all patients. Given the prevalence of nutritional risks, the treatment of lean muscle mass loss remains a challenge in clinical practice. For this reason, a multidisciplinary approach with targeted nutritional therapy is crucial to improve the quality of care in oncology. A protein level of 1-1.2 g/kg bw is suggested for the maintenance of muscle mass.However, it has been shown that this amount is not sufficient to support ALM in patients with tumor diseases. Only an amount above 1.4 g/kg bw has been associated with a positive effect on muscle mass. Adequate dietary protein intake is essential for the maintenance of numerous physiological processes, including muscle protein synthesis and muscle function. Sufficient energy and protein intake is necessary to support muscle protein synthesis. The scientific literature frequently discusses the relationship between daily protein intake and its distribution over the main meals. The evening meal is particularly important for the maintenance of ALM.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent
* At least 45 years of age
* Sufficient knowledge of the German language
* Indication to undergo radio(chemo)therapy with at least 10 fractions

Exclusion Criteria:

* Participation in other interventional studies
* Pregnancy/breastfeeding
* Previous intake of high-calorie supplementary food or intravenous nutrition
* BMI < 18.5
* When performing the bioimpedance measurement: patients with pacemakers, defibrillators and other implanted automatic devices

Ages: 45 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Indication for radio(chemo)therapy in the presence of one of the following histologically confirmed tumor diseases: Thorax, head and neck, breast, abdomen/pelvis, brain, bone metastases, prostate
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Protein uptake in g/kg body weight | baseline, end of radiotherapy and 3 months after Radiotherapy
  Change in the amount of protein consumed and its distribution over the main meals by means of a dietary questionnaire before, at the end and 3 months after completion of radiotherapy.

SECONDARY OUTCOMES:
Weight in kg | baseline, end of radiotherapy and 3 months after Radiotherapy
  Body Weight
Muscle mass in kg | baseline, end of radiotherapy and 3 months after Radiotherapy
  Evaluation of Muscle mass via Bioimpedance Measurements
Quality of Life (EORTC QLQ C30) in 5-tier likert scale (higher scores = better) | baseline, end of radiotherapy and 3 months after Radiotherapy
  Health Related Quality of Life with EORTC QLQ C30
Height in m | baseline, end of radiotherapy and 3 months after Radiotherapy
  Height
Fatigue in 5-tier likert scale (higher scores = worse) | baseline, end of radiotherapy and 3 months after Radiotherapy
  FACIT F Questionnaire
BMI in kg/m² | baseline, end of radiotherapy and 3 months after Radiotherapy
  BMI calculated from weight and Hight
Treatment Toxicity via CTCA criteria (5 tier scale; higher = worse) | baseline, weekly during radiotherapy, end of treatment, follow up (up to 1 year, on average every 3 months)
  Common Terminology Criteria for Adverse Events (CTCAE) version 5
Treatment Toxicity via PROMs (5 tier scale; higher = worse) | baseline, weekly during radiotherapy, end of treatment, follow up (up to 1 year, on average every 3 months)
  Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine Berlin, Berlin, State of Berlin, Germany